CLINICAL TRIAL: NCT06040099
Title: Phase II Single-Arm Study of Durvalumab and Bevacizumab Following Transarterial Radioembolization Using Yttrium-90 Glass Microspheres (TheraSphere™) in Unresectable Hepatocellular Carcinoma Amenable to Locoregional Therapy
Brief Title: A US Study to Evaluate Transarterial Radioembolization (TARE) in Combination With Durvalumab and Bevacizumab Therapy in People With Unresectable Hepatocellular Carcinoma Amenable to TARE
Acronym: EMERALD-Y90
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D933GC00002
Record Dates: First submitted 2023-09-11; First posted 2023-09-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: TARE; Durvalumab; Bevacizumab; Liver Cancer; Y90
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — durvalumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Yttrium 90 glass microspheres TARE in combination with Durvalumab and Bevacizumab (Experimental): Participants will undergo Yttrium 90 glass microspheres TARE according to the dosimetry recommendation.
  Interventions: Drug: Durvalumab; Drug: Bevacizumab; Procedure: Transarterial Radioembolization (TARE)

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous)
  Other Names: MEDI4736, IMFINZI
Drug: Bevacizumab — Bevacizumab IV (intravenous)
  Other Names: AVASTIN, ZIRABEV
Procedure: Transarterial Radioembolization (TARE) — Yttrium 90 glass microspheres will be administered
  Other Names: TheraSphere

SUMMARY:
The purpose of this study is to measure the efficacy and safety of durvalumab intravenous (IV) solution plus bevacizumab IV solution after transarterial radioembolization (Yttrium 90 glass microspheres TARE) in participants with unresectable hepatocellular carcinoma (HCC) amenable to embolization.

DETAILED DESCRIPTION:
A Phase II single-arm study conducted in participants with unresectable Hepatocellular carcinoma (HCC) eligible for embolization and not eligible for or who have declined treatment with resection and/or ablation or liver transplant.

Participants with previous Transarterial Chemoembolization (TACE) or TARE associated with the curative setting are permitted with a 6-month washout.

Approximately 120 participants with unresectable but amenable to locoregional therapy HCC eligible for embolization will be screened in the study at approximately 20 sites in the US to enroll approximately 60 participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with confirmed unresectable HCC
* Participants with Lung dose threshold for Yttrium 90 glass microspheres of 30 Gy (equal or less than 30 Gy per treatment for glass) and an estimated Future liver remnant volume (FLRV) ≥ 30% of whole liver volume.
* Participants with more than 1 prior embolization are permitted if more than 12 months ago, for a different primary lesion, and FLR > 30%.
* Participants with no evidence of extrahepatic disease on any available imaging
* Participants with one or more measurable lesions, unilobar disease for participants with segmental or right anterior/posterior portal vein invasion (Vp1/Vp2) and eligible for Yttrium 90 glass microspheres TARE.
* Participants having Child-Pugh score class A.
* Participants having ECOG performance status of 0 or 1 at enrollment
* Adequate organ and marrow function

Exclusion Criteria:

* Disease amenable to curative surgery, ablation or transplantation. Transplant patients are considered eligible if outside of Milan criteria and not currently listed for transplant.
* Participants co-infected with HBV and HDV
* Any history of nephrotic or nephritic syndrome.
* Clinically significant (eg, active) cardiovascular disease
* Participants with uncontrolled hypertension
* History of hepatic encephalopathy
* Known hereditary predisposition to bleeding or thrombosis; any prior or current evidence of bleeding diathesis.
* Receipt of more than 1 prior embolization (TACE or TARE) treatment/procedure
* Participant has received any prior anticancer systemic therapy for unresectable HCC.
* History of arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to enrollment.
* History of abdominal fistula or gastrointestinal (GI) perforation, non-healed gastric ulcer that is refractory to treatment, or active GI bleeding within 6 months prior to enrollment

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2027-01-13 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From Day 1 until date of progressive disease or death [Approximately 3 years]
  PFS is defined as the time from Day 1 (day of TARE) until the date of progressive disease per modified Response Evaluation Criteria in Solid Tumors (mRECIST), as assessed by the investigator, or death due to any cause. It is measured to assess the efficacy of TARE followed by durvalumab monotherapy followed by durvalumab + bevacizumab in participants with unresectable HCC amenable to locoregional therapy.

SECONDARY OUTCOMES:
Number of participants with Adverse events (AEs) | From Screening (Day -28 to Day 1) until 90 days after the last dose of study drug
  To assess the safety of the sequence of TARE followed by durvalumab monotherapy followed by durvalumab + bevacizumab in participants with unresectable HCC amenable to locoregional therapy
Objective Response Rate (ORR) | From Day 1 until progression, or the last evaluable assessment in the absence of progression (Approximately 3 years)
  ORR is defined as the proportion of participants who have a confirmed complete response or partial response, as determined by the investigator per mRECIST. It is assessed after TARE followed by durvalumab monotherapy followed by durvalumab + bevacizumab in participants with unresectable HCC amenable to locoregional therapy.
Overall Survival (OS) | Day 1 to 18 months or until death (Approximately 3 years)
  OS is defined as the time from the start of TARE until the date of death due to any cause. It is assessed after TARE followed by durvalumab monotherapy followed by durvalumab + bevacizumab in participants with unresectable HCC amenable to locoregional therapy.
Duration of Response (DoR) | Time from first documented response until documented progression (Approximately 3 years)
  DoR is defined as the time from the date of first documented response (that is subsequently confirmed) until the date of documented progression per mRECIST as assessed by the investigator, or death due to any cause. It is assessed after TARE followed by durvalumab monotherapy followed by durvalumab + bevacizumab in participants with unresectable HCC amenable to locoregional therapy.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Research Site, Aurora, Colorado
  - Research Site, Gainesville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Trenton, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home